CLINICAL TRIAL: NCT07186764
Title: Evaluation of the Overall Quality of Life and Gynecological Follow-up of Patients Treated for Mayer-Rokitansky-Küster-Hauser (MRKH) Syndrome at the Toulouse University Hospital
Brief Title: Evaluation of the Quality of Life and Gynecological Follow-up of Patients Treated for Mayer-Rokitansky-Küster-Hauser (MRKH) Syndrome
Acronym: MOQA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/25/0251; ID-RCB (Other: 2025-A01148-41)
Record Dates: First submitted 2025-09-03; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mrkh Syndrome
Keywords: MRKH; Mayer-Rokitansky-Küster-Hauser; gynecology; vaginal aplasia; quality of life; MRKH syndrome
MeSH Terms: conditions — Mullerian aplasia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Mayer-Rokitansky-Küster-Hauser (MRKH) syndrome: Women patients with Mayer-Rokitansky-Küster-Hauser syndrome
  Interventions: Other: Questionnaires; Other: Semi-directed interview
- Control group: patients followed in the gynecology department but not suffering from Mayer-Rokitansky-Küster-Hauser syndrome
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — questionnaires: WHOQOL-BREF (Quality of Life Study Questionnaire), FSFI (Female Sexual Function Index), FSDS-R (The Femala sexual distress scale-revised), Rosenberg scale (self-esteem assessment)
Other: Semi-directed interview — Semi-directed interview on the treatment pathway and the impact of utero-vaginal aplasia on intimate and personal life
  Groups: Patients with Mayer-Rokitansky-Küster-Hauser (MRKH) syndrome

SUMMARY:
Mayer-Rokitansky-Küster-Hauser (MRKH) syndrome affects 1 in 4,500 women and consists of utero-vaginal aplasia in 46 chromosom XX women, most often diagnosed in the presence of primary amenorrhea. This diagnosis, occurring in adolescence during the period of identity formation, can have significant psychological repercussions. This malformation can alter the body image and personal relationships of affected patients, beyond the impact on their sexual lives. Management around the disclosure is a crucial moment for these patients. Individual or group psychological support is systematically offered.

Several international studies show that these patients experience a decline in their quality of life, and they are more anxious and depressed. Participation in support groups improves this state.

The objective of this study is therefore to better understand Mayer-Rokitansky-Küster-Hauser (MRKH) syndrome and the issues patients may face. For this reason, it seems essential to us to evaluate the overall quality of life, the quality of sexual life, the psychological state and the gynecological follow-up of women before or after treatment for vaginal aplasia.

DETAILED DESCRIPTION:
Mayer-Rokitansky-Küster-Hauser (MRKH) syndrome affects 1 in 4,500 women. In its classic form, it consists of uterovaginal aplasia in 46XX chromosom women, most often diagnosed in the presence of primary amenorrhea. This diagnosis, occurring in adolescence during the period of identity formation, can have significant psychological repercussions. Indeed, this uterovaginal aplasia is responsible for the inability to achieve vaginal penetration during sexual intercourse, the absence of menstruation, and the inability to conceive.

It is therefore easy to understand that this malformation can alter the body image and personal relationships of affected patients, beyond the impact on their sexual lives. Management around the time of disclosure is a crucial moment for these patients. Individual or group psychological support is systematically offered.

Before the 2010s, surgical techniques for vaginal creation were widely proposed, which was rejected in uterine transplant research protocols. Since 2014 (the first uterine transplant), expert physicians working with the Rare Gynecological Pathology Reference Centers have offered patients who wish to undergo vaginal self-dilation (the Frank technique). This neovagina allows for sexual intercourse with vaginal penetration. It is also an essential prerequisite in uterine transplant protocols, the criterion for which is a vaginal depth greater than 7 cm.

This condition requires a multidisciplinary approach. The discovery of this malformation raises many questions, due to the significant social, legal, and ethical implications: What do these patients think of their overall quality of life and their sexual quality? Do they have more psychological disorders than the general population? Are they well-monitored gynecologically? Does the treatment of utero-vaginal aplasia improve patients' quality of life? Several international studies show that these patients experience a decline in their quality of life; they are more anxious and more depressed. Participation in support groups improves this condition. These are older studies with cohorts of patients who most often benefited from surgical treatment, which is no longer the standard method today. These studies therefore do not allow an assessment of the current population.

The objective of this study is therefore to better understand Mayer-Rokitansky-Küster-Hauser (MRKH) syndrome and the issues patients may face. To this end, we believe it is essential to assess the overall quality of life, sexual quality, psychological state, and gynecological follow-up of women before or after treatment for vaginal aplasia. Indeed, women must be able to fully experience their sexuality and achieve fulfillment through it. The impact of proposed medical treatments on sexuality must therefore be a concern for practitioners.

The evaluation of functional outcomes and the potential impact of our treatments must therefore be an integral part of follow-up.

Currently, there is little data regarding long-term outcomes after medical or surgical treatment.

The objective is to identify areas for improvement which could bring to the management and follow-up of this syndrome, in order to subsequently offer a personalized care pathway and better meet the needs of patients.

ELIGIBILITY:
Inclusion Criteria:

* For Mayer-Rokitansky-Küster-Hauser patients:

  * Patient over 18 and under 50
  * Confirmed diagnosis of Mayer-Rokitansky-Küster-Hauser syndrome
  * Diagnosis announced more than 1 year ago
  * Patient treated by the CRMR PGR
  * Patient affiliated with or benefiting from a social security scheme
  * Fluency in French
* For the control population:

  * Patient over 18 and under 50
  * Patient affiliated with or benefiting from a social security scheme
  * Fluency in French

Exclusion Criteria:

* For Mayer-Rokitansky-Küster-Hauser patients:

  * Minors over 50 years of age
  * Recent diagnosis < 1 year
  * Other causes of uterine or vaginal aplasia, surgical or congenital

    • Patients benefiting from a legal protection measure (guardianship, curatorship, legal protection)
  * Patients unable to understand or answer the questionnaires
* For the control population:

  * Minors over 50 years of age
  * Patients benefiting from a legal protection measure (guardianship, curatorship, legal protection)
  * Patients unable to understand or answer the questionnaires

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with Mayer-Rokitansky-Küster-Hauser syndrome and patients followed in gynecological consultation without the presence of this syndrome
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the overall quality of life of patients with Mayer-Rokitansky-Küster-Hauser syndrome. | One hour after the inclusion
  Comparison of the score obtained on the WHOQOL BREF questionnaire between women with Mayer-Rokitansky-Küster-Hauser syndrome and the control population (score from 0 to 100, 0 corresponding to the worst quality of life and 100 to the best possible quality of life)

SECONDARY OUTCOMES:
Evaluation of the quality of sexual life | 1 hour after the inclusion
  FSFI questionnaire response score (Female sexual function Index). A total score of 26.55 has been proposed as a cut-off value for the diagnosis of sexual dysfunction, with the maximum score being 36
Assessment of distress regarding sexuality | 1 hour after the inclusion
  Female Sexual Distress Scale-Revised (FSDS-R) questionnaire response score. A score > 15 indicates distress related to dysfunctional symptoms and therefore sexual dysfunction. The response to the first question is the best reflection of sexual distress.
Self-esteem assessment | 1 hour after the inclusion
  Response score to the Rosenberg Self-Esteem Scale questionnaire. Score obtained between 10 and 40, a score <25 indicates very low self-esteem, and a score >39 corresponds to high self-esteem
Evaluation of gynecological monitoring of patients | 1 hour after the inclusion
  existence or not of regular gynecological monitoring
Qualitative evaluation of the impact of utero-vaginal aplasia on intimate life | 1 hour after the inclusion
  questions asked during the semi-directed interview in patients with Mayer-Rokitansky-Küster-Hauser syndrome
Evaluation of the functional impact of the treatment | 1 hour after the inclusion
  The patient will be asked to participate in a semi-structured interview consisting of questions designed to analyze the impact of the condition and its treatment on the life experiences of women with Mayer-Rokitansky-Küster-Hauser syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Endocrino-gynéco-pédiatrie, Hôpital des Enfants, 330 Avenue de Grande Bretagne, Toulouse, France

IPD SHARING:
Plan to Share IPD: No